CLINICAL TRIAL: NCT03459625
Title: Mindfulness and Parent Stress Reduction: Improving Outcomes for Children With Autism Spectrum Disorder
Brief Title: Mindfulness for Parents of Children With Autism Spectrum Disorder Autism Spectrum Disorder
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: California State University, Fullerton (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cameron Neece, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5110264
Record Dates: First submitted 2018-02-28; First posted 2018-03-09 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized controlled trial of 138 families that will be conducted in three cohorts. Each cohort will involve a recruitment phase of 46 participants. Within each cohort parents will be randomly assigned to the MBSR (N=23) or PE group (N=23), and the groups will run concurrently.
Who Masked: Outcomes Assessor
Masking Description: Participants will participate in laboratory assessments at baseline and immediately post-treatment, as well as at 6 months and 12 months post-treatment. Measures include standardized and validated parent and teacher questionnaires, gold-standard psychological assessments, and observational and interview ratings. All assessors for laboratory assessments will remain blind to treatment group assignment for the duration of the project. Teachers will also be blind to treatment group assignment. Research assistants involved in observational coding will be blind to both treatment condition and visit time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (MSBR) (Experimental): MSBR (Kabat-Zinn, 1990), 8-week group-based intervention where participants learn mindfulness skills to help alleviate parenting stress among parents of young children with Autism Spectrum Disorder.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MSBR)
- Psychoeducational Support Group (PE) (Active Comparator): PE is a 8-week group-based intervention to provide psychosocial support and resources for parents of young children with Autism Spectrum Disorder.
  Interventions: Behavioral: Psychoeducational Support Group (PE)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MSBR) — MBSR includes eight weekly 2.5-hour group sessions, a day-long (6hr) meditation retreat on the weekend during week six, 45 minutes of daily home practice guided by instructional audio CDs, and an MBSR parent workbook. Formal mindfulness exercises aim to increase the capacity for mindfulness and include a body scan, mindful yoga, and sitting meditation. Participants are also taught to practice mindfulness informally in everyday activities. In session, didactic instruction on stress physiology and using mindfulness for coping with stress in daily life is provided. Participants practice formal mindfulness exercises, break into dyads to discuss their daily homework practice, and meet as a larger group to ask questions related to the practice of mindfulness in everyday life.
  Arms: Mindfulness-Based Stress Reduction (MSBR)
Behavioral: Psychoeducational Support Group (PE) — The PE consists of 8-weekly 2.5-hour sessions, a day-long (6hr) Family Resource Fair during week six, daily homework that includes monitoring progress on goals identified at the end of each session, and a workbook for parents of children with special needs that provides parents with information regarding their child's development, disability, and associated considerations. Weekly topics for discussion include Preparing for Individualized Education Plan (IEP) meetings, Communicating with Teachers, Advocacy, Sibling Issues, and Community Resources.
  Arms: Psychoeducational Support Group (PE)

SUMMARY:
The current study examines the efficacy of Mindfulness-Based Stress Reduction (MBSR) to reduce parenting stress, lessen parental reactivity and negativity, and decrease child externalizing behaviors among families of children with Autism Spectrum Disorder (ASD). The design is a randomized controlled trial of 138 families of preschool-aged children with ASD. Parents of children with ASD will be randomized to MBSR or to a Psychoeducational (PE) support control group matched for clinical contact and dosage (see details on interventions below). Families will participate in laboratory assessments at baseline and immediately post-treatment, as well as at 6 months and 12 months post-treatment. Measures include standardized and validated parent and teacher questionnaires, gold-standard psychological assessments, and observational and interview ratings.

DETAILED DESCRIPTION:
Families of children with Autism Spectrum Disorder (ASD) experience heightened risk due to elevated rates of clinically-significant parenting stress and child externalizing behavior problems. Parenting stress is a robust predictor of subsequent externalizing challenges in children with ASD. Nonetheless, few evidenced-based treatments exist for reducing parenting stress in these families. The mechanisms through which parenting stress influence child externalizing problems are also unclear, although preliminary evidence suggests the potential role of negative parenting behaviors. This study comprehensively addresses these considerations by testing the efficacy of Mindfulness-Based Stress Reduction (MBSR) as an intervention to reduce parenting stress, lessen parental reactivity and negativity, and decrease child externalizing behaviors.

MBSR is particularly well-suited for parents of children with ASD given the intervention emphasis on teaching participants to manage reactivity in the context of persistent stress. However, the efficacy of MBSR has yet to be established for this population. The present investigation extends preliminary investigations of mindfulness approaches by: 1) conducting a stringent test of MSBR using an active psychoeducational (PE) control, 2) developing population-specific content and testing the efficacy of MSBR for parents of children with ASD, 3) utilizing a highly diverse, underserved community-based sample, 4) examining the mechanisms underlying observed treatment effects, and 5) employing multi-method longitudinal measurement from multiple sources in order to examine immediate and long-term treatment effects.

The current study is a randomized controlled trial of 138 families of preschool-aged children with ASD. Parents will be randomized to MBSR or to a PE support group matched for clinical contact and dosage. Families will participate in laboratory assessments at baseline and immediately post-treatment, as well as at 6 months and 12 months post-treatment. Measures include standardized and validated parent and teacher questionnaires, gold-standard psychological assessments, and observational and interview ratings.

The MBSR intervention includes eight weekly 2.5-hour group sessions, a day-long (6hr) meditation retreat on the weekend during week six, 45 minutes of daily home practice guided by instructional audio CDs (portable CD players will be provided when necessary), and an MBSR parent workbook. Formal mindfulness exercises aim to increase the capacity for mindfulness (present-moment awareness with a compassionate, non-judgmental stance) and include a body scan, mindful yoga, and sitting meditation. Participants are also taught to practice mindfulness informally in everyday activities. In session, didactic instruction on stress physiology and using mindfulness for coping with stress in daily life is provided. Participants practice formal mindfulness exercises, break into dyads to discuss their daily homework practice, and meet as a larger group to ask questions related to the practice of mindfulness in everyday life.

In order to provide a rigorous test of the contributions of mindfulness techniques, the current investigation will control for therapeutic effects associated with clinician contact and group support by comparing MBSR to a PE support condition matched for dosage. The PE condition also consists of 8-weekly 2.5-hour sessions, a day-long (6hr) Family Resource Fair during week six (wherein families will attend talks by professionals, explore available local resources, and meet with service providers), daily homework that includes monitoring progress on goals identified at the end of each session, and a workbook for parents of children with special needs that provides parents with information regarding their child's development, disability, and associated considerations.

Establishing an efficacious stress reduction intervention to target mechanisms linking parenting stress, negative parenting behaviors, and child externalizing problems will advance clinical science and optimize outcomes for children with ASD and their families.

ELIGIBILITY:
Inclusion Criteria:

* Child community diagnosis of ASD confirmed by study administered assessments
* Age 3 to 5 years
* Elevated parenting stress as indexed by a total score above the recommended cutoff at the 85th percentile on the Parenting Stress Index-4 (Abidin, 1995)
* Abbreviated Battery IQ (ABIQ) score above 35 on the Stanford-Binet Intelligence Scales 5th Edition ABIQ to ensure task validity (SB5 ABIQ; Roid, 2003)

Exclusion Criteria:

* Positive screen for active parental psychosis, substance abuse, or suicidality according to the associated modules of the Structured Clinical Interview for DSM Disorders, SCID, Research Version Non-Patient Edition (First, Spitzer, Gibbon, & Williams, 2002)
* Parent participation in an auxiliary mental health treatment or support group
* < 3 years or > 5 years of age

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron L Neece, Ph.D., Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Protocol Enrollment (118) reflects the number of parent participants. The Total Started in Participant Flow (118) reflects the number of parent participants who were enrolled and assigned to each arm. Of note, one participant dropped out of the study and requested to not have their data used/reported. Thus, the total sample we report is N=117
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Started | 60 | 58
Completed | 59 | 58
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE) | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Customized [Mean (Standard Deviation); unit: years] | 34.56 (7.541) | 34.67 (7.529) | 34.61 (7.535)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject withdrew consent prior to data analysis
  Participants
    Female | 13 | 10 | 23
    Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 28 | 60
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Child Externalizing Behavior Problems as Evidenced by Reductions in the Externalizing Scores on a Standardized Parent-report Questionnaire.
Description: Assessment will be based on reductions parent ratings on the Externalizing Problems t-score of the Child Behavior Checklist-Ages 1.5-5. The Child Behavior Checklist has 99 items that assess the degree or frequency of child behavior problems. Each item is rated on a scale of 0 (not true), 1 (somewhat or sometimes true), or 2 (very true or often true). T-scores on the Externalizing Problems sub-scale of the Child Behavior Checklist have a theoretical population mean of 50 and a standard deviation of 10. Higher scores indicating more behavior problems. A t-score between 60 and 63 on the Externalizing Problems sub-scale is considered Borderline and a t-score above 63 is considered Clinical.
Time Frame: At baseline
Population: All study participants are parents of children ages 3 to 5 years with diagnosis of Autism Spectrum Disorder confirmed by study administered assessments. These participants were drawn from the Inland Empire region of Southern California.
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
t-scores | 68.40 (11.335) | 66.49 (11.393)

2. Primary Outcome: Child Externalizing Behavior Problems as Evidenced by Reductions in the Externalizing Score on a Standardized Parent-report Questionnaire.
Description: as for outcome 1
Time Frame: Within 4 weeks of completing last intervention session (session 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 61.64 (11.704) | 62.82 (10.878)

3. Primary Outcome: Child Externalizing Behavior Problems as Evidenced by Reductions in the Externalizing Score on a Standardized Parent-report Questionnaire.
Description: as for outcome 1
Time Frame: 6-month follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 61.69 (12.148) | 64.07 (9.773)

4. Primary Outcome: Child Externalizing Behavior Problems as Evidenced by Reductions in the Externalizing Score on a Standardized Parent-report Questionnaire.
Description: as for outcome 1
Time Frame: 12-month follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 62.03 (12.388) | 65.50 (9.538)

5. Secondary Outcome: Parenting Stress
Description: Assessment will be based in parent participant reports on the Parental Distress sub-scale of the Parenting Stress Index-Fourth Edition, Short Form. The Parenting Stress Index includes 36 items that are rated on a five-point scale that ranges from 1 (strongly agree) to 5 (strongly disagree). Scores on the Parental Distress sub-scale of the Parenting Stress Index-Fourth Edition, Short Form range from 12 to 60, with higher scores indicating more parental distress.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 37.4717 (9.19156) | 37.4340 (8.35397)

6. Secondary Outcome: Parenting Stress
Description: as for outcome 5
Time Frame: Within 4 weeks of completing last intervention session (session 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 28.8000 (9.44132) | 33.1739 (7.17187)

7. Secondary Outcome: Parenting Stress
Description: as for outcome 5
Time Frame: 6-month follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 27.9615 (10.12514) | 32.1333 (7.78032)

8. Secondary Outcome: Parenting Stress
Description: as for outcome 5
Time Frame: 12-month follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
Number analyzed (Participants) | 59 | 58
units on a scale | 26.0323 (9.23935) | 32.6154 (6.87067)

ADVERSE EVENTS:
Time Frame: 3 years, 11 months
Arm/Group | Mindfulness-Based Stress Reduction (MSBR) | Psychoeducational Support Group (PE)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58

LIMITATIONS AND CAVEATS:
The onset of the COVID-19 pandemic and associated restrictions on in-person activities changed our procedures mid-study and likely impacted parents' stress levels and experiences in the interventions. Additionally, while the use of an active comparator was a significant strength of the study's design, we did not have a no-intervention control group and therefore we cannot evaluate the benefit of the MSBR of PE interventions relative to normative changes in parenting stress over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03459625/Prot_SAP_ICF_000.pdf